CLINICAL TRIAL: NCT02123693
Title: The Role of Osteopathic Treatment in the Axial Variations of the Lumbar Spine: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DYNOST-01
Record Dates: First submitted 2014-04-24; First posted 2014-04-25 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Low Back Pain
Keywords: Osteopathic manipulative treatment; Low back pain; Dynamic MRI
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Osteopathic Manipulative Treatment (Experimental): 5 sessions of treatment will be carried out: the first 3 weekly, and the remaining 2 after 15 days. The type of treatment will be based on indirect techniques
  Interventions: Other: Osteopathic manipulative treatment
- Sham therapy (Sham Comparator): 5 sessions of treatment will be carried out: the first 3 weekly, and the remaining 2 after 15 days. The type of treatment will be based on specific parameters set out previously based on a predetermined protocol
  Interventions: Other: Sham Therapy
- No intervention (Other): Patients in this group will not receive any type of intervention, both therapeutic than fictitious, and will not be evaluated by any operator
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: Osteopathic manipulative treatment
  Arms: Osteopathic Manipulative Treatment
Other: Sham Therapy
  Arms: Sham therapy
Other: No Intervention
  Arms: No intervention

SUMMARY:
The aim of the present study is to determine whether there is a relationship between osteopathic treatment and the change of physiological axes of the lumbar spine, through the use of Dynamic Magnetic Resonance Imaging.

ELIGIBILITY:
Inclusion Criteria:

* will be admitted patients of both genders
* patients with chronic low back pain at baseline
* patients aged between 18 and 35 years

Exclusion Criteria:

* patients diagnosed with the disease of the musculoskeletal system or congenital malformation of the column
* patients with disorders of the pelvic floor, or who have undergone surgery of the reproductive system
* patients with neurological disorders that can cause painful symptoms of lumbar segment

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Baseline changes in degree of flection of lumbar spine | at entry and after 8 weeks

SECONDARY OUTCOMES:
Baseline changes in Visual Analogue Scale | at entry and after 8 weeks
Baseline changes in Roland-Morris questionnaire | at entry and after 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Radiology Unit II, University Hospital San Salvatore L'Aquila, L’Aquila, Abruzzo, Italy